CLINICAL TRIAL: NCT05177172
Title: Synergistic Effect of Oat Beta-glucans and Oat Polar Lipids on Postprandial Glucose Response
Brief Title: Effect of Oat Compounds on Postprandial Glucose Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Anne Nilsson, Associate professor, Lund University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Scanoats
Record Dates: First submitted 2021-12-01; First posted 2022-01-04 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Healthy Subjects
Keywords: Prevention; food; diabetes type 2; postprandial glucose regulation; appetite; oat; polar lipids; obesity; glucose tolerance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Gyrate Atrophy; Obesity

STUDY DESIGN:
Intervention Model Description: Randomised food study in healthy subjects
Who Masked: Participant
Masking Description: Four test products and one reference product (control). Participants are not aware of which product that is served at each visits
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control (Placebo Comparator): White wheat flour bread
  Interventions: Other: Control
- High betaglucans (Experimental): White wheat flour bread included beta glucans with the highest amounts in this study
  Interventions: Other: High beta glucans
- Low beta glucans (Experimental): White wheat flour bread included beta glucans with the lowest amounts in this study
  Interventions: Other: Low beta glucans
- Low beta glucans + low polar lipids (Experimental): White wheat flour bread included a combination of the lowest amounts of beta glucans and polar lipids
  Interventions: Other: Low beta glucans + low polar lipids
- low polar lipids (Experimental): White wheat flour bread included polar lipids
  Interventions: Other: Polar lipids

INTERVENTIONS:
Other: High beta glucans — higher dose betaglucans
  Arms: High betaglucans
Other: Low beta glucans — lower dose beta glucans
  Arms: Low beta glucans
Other: Low beta glucans + low polar lipids — low dose betaglucans in a combination with low dose of polar lipids
  Arms: Low beta glucans + low polar lipids
Other: Polar lipids — low dose polar lipids
  Arms: low polar lipids
Other: Control — No beta glucans or polar lipids
  Arms: Control

SUMMARY:
In this project we will investigate synergistic effects of oat polar lipids and beta glucans on postprandial glucose tolerance

ELIGIBILITY:
Inclusion Criteria:

* healthy
* BMI 20-28 kg/m2
* Diet which follows the Nordic Nutrition Recommendations (non-vegetarian)

Exclusion Criteria:

* fasting glucose > 6.1 mmol/L
* metabolic diseases
* gastrointestinal disease
* chronic and/or psychological disease
* food allergy
* Vegetarian or vegan diets, or other special diets

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-01-19 (Actual); Study Completion 2022-01-19 (Actual)

PRIMARY OUTCOMES:
Glucose tolerance | 3 hours. Fasting (time =0 minutes), 15 minutes, 30 minutes, 45 minutes, 60 minutes, 90 minutes, 120 minutes, 150 minutes, 180 minutes
  Postprandial glucose concentrations (mmol/L). The incremental area under the curve will be calculated and expressed as mmol*minutes/litre.

SECONDARY OUTCOMES:
Subjective appetite variables | 3 hours. Fasting (time =0 minutes), 15 minutes, 30 minutes, 45 minutes, 60 minutes, 90 minutes, 120 minutes, 150 minutes, 180 minutes
  Postprandial sensation of hunger, satiety, and desire to eat will be determined with a 100 millimeter visual analogue scale (VAS). The left end of the VAS scale represent "not at all" (e.g. hungry) and right end of the scale represented "extremely". One scale for each parameter will be used. The total area under the curve will be calculated, and the results will be expressed as millimeter*minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Lund University, Food Technology, Engineering and Nutrition, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Will be available after request